CLINICAL TRIAL: NCT06625268
Title: Machbarkeit Und Explorative Validierung Des PA-100-AST-Systems Bei Frauen Mit Verdacht Auf Eine Unkomplizierte Harnwergsinfektion in Der Hausarztpraxis - Eine Pilotstudie
Brief Title: Rapid Point-of-care Bacteriuria and Microbial Susceptibility for Women With Suspected Uncomplicated Urinary Tract Infections: Diagnostic Accuracy in General Practice.
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-3379-BO
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Urinary Tract Infection (Diagnosis)
Keywords: urinary tract infection; women; general practice; diagnosis; primary care; point-of-care test
MeSH Terms: conditions — Urinary Tract Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with suspected UTI: Adult women with suspected uncomplicated urinary tract infections

SUMMARY:
In this study, adult women presenting at their general practitioner with a likely bladder infection (with symptoms like a burning sensation when urinating, pain in the lower abdomen, and frequent or urgent need to urinate) will be invited. After informed consent, women provide a urine sample, which is tested using a new system called the PA-100-AST (from the manufacturer Sysmex). This point-of-care test showed first evidence to be able to quickly detect the presence of bacteria commonly responsible for bladder infections. If bacteria are found, the test also checks which antibiotics may work best to treat the infection. Additionally, a sample of the urine is sent to a lab for a traditional culture test, which is considered the most accurate method. The goal of this study is to compare the accuracy of the PA-100-AST system to the lab-based test to see how well it works in general practice.

DETAILED DESCRIPTION:
The PA-100-AST urine analyzer from Sysmex is a rapid point-of-care test currently registered as a medicinal product. The system identifies bacteriuria (≥ 50,000 CFU/mL) and reports antibiotic susceptibility results as susceptible (S), susceptible with increased exposure (I), resistant (R), or not applicable (NA) for amoxicillin/clavulanic acid, ciprofloxacin, fosfomycin, nitrofurantoin, and trimethoprim, based on EUCAST standards. Although the system detects bacteriuria, it does not inform the user of the specific bacterial species involved, providing only a positive or negative result.

The PA-100 cartridge is designed to detect common uropathogens: Escherichia coli, Klebsiella pneumoniae, Proteus mirabilis, Enterococcus faecalis, and Staphylococcus saprophyticus. A proprietary internal algorithm classifies bacteria into one of three groups (Enterobacterales, Staphylococcus, or Enterococcus) and applies appropriate EUCAST breakpoints.

This product is authorized and CE-marked in the European Union for point-of-care use in women with suspected uncomplicated urinary tract infections (UTIs).

However, the PA-100-AST system has not yet been evaluated in a general practice setting. The goal of this study is to compare the results of the Sysmex PA-100-AST with laboratory-based urine culture in a consecutive sample of adult women recruited from general practices.

Recruitment. Adult, non-pregnant women with symptoms suggestive of uncomplicated UTI will be recruited consecutively and prospectively during routine consultations in at least four general practices across two German practice-based research networks (Bavaria and Thuringia). Informed consent will be obtained from all participants.

Outcomes. The primary outcome measure is diagnostic accuracy compared with urine culture. Urine culture positivity is defined as a bacterial count of at least 50,000 CFU/ml (per the instructions for use) of one of the species detected by the PA-100-AST (index test). Additionally, the diagnostic accuracy of the index test will be assessed against varying thresholds for urine culture positivity (from 1,000 to 100,000 CFU/ml or greater).

Another key outcome is the agreement between the susceptibility test results from the index test and the reference laboratory-based susceptibility test. Exploratory subgroup analyses will include assessments based on age, dipstick test results, and symptom severity at presentation.

Data Collection. The index test will be conducted immediately after enrolment on fresh urine (within 30 minutes of collection). A pragmatic approach will be followed, with microbiological analysis carried out by the laboratories that typically serve the participating practices. These laboratories adhere to common quality standards according to the German laboratory guidelines (Harnwegsinfektionen: Qualitätsstandards in der mikrobiologisch-infektiologischen Diagnostik, MIQ-02) and apply EUCAST criteria for susceptibility testing. According to STARD recommendations, clinicians performing the index test, as well as laboratory technicians and microbiologists conducting the urine culture, are blinded to the results of each other´s tests. Clinical data are collected using a validated patient questionnaire at the initial presentation, and management decisions are recorded during routine consultation. Dipstick test results are measured through Combur test stripes (Roche Diagnostics).

Data Analysis. Descriptive statistics will be presented using appropriate summary measures such as mean (SD), median (IQR), and absolute and relative frequencies.

Diagnostic accuracy measures (sensitivity, specificity, predictive values, and likelihood ratios) will be reported with corresponding 95% confidence intervals.

Kappa coefficients and corresponding statistical tests will be used to assess agreement between categorical variables (with statistical significance set at p less than 0.05) for susceptibility test results.

Sample Size. The initial sample size calculation assumed a sensitivity of 98.8% and specificity of 98.4% based on manufacturer data. Given a prevalence of 70%, we estimated that 101 patients would be required to estimate specificity, and 51 patients to estimate sensitivity, with a 95% confidence interval (CI) width of 0.1. However, after the protocol was approved, a clinical evaluation in a hospital setting (PMID: 38825624) was published, reporting a sensitivity of 84% and a specificity of 99.4% for the PA-100-AST, using a threshold of 50,000 CFU/ml as per the instructions for use. Given the more realistic estimates from this study, the sample size was recalculated. Based on the revised sensitivity and specificity estimates, and a 50,000 CFU/ml culture positivity threshold for which a decreased prevalence from 0.70 to 0.60 can be expected, the required sample size increased from 101 to 345 participants. Due to no project-specific funding, and in agreement with the sponsor, this was deemed unfeasible. Therefore, the aim to recruit 200 participants, which, under the assumption outlined above, will result in a 95%CI width of 0.13 instead of the initially planned width of 0.1.

Role of manufacturer. This study is investigator-initiated. Sysmex has provided the urine analyzer free of charge but has no involvement in the study design, implementation (aside from supplying detailed instructions for use as well as technical assistance), data preparation, analysis, interpretation, or publication of results. None of the investigators receive any funding or benefits from Sysmex or other device manufacturers.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 18 or older
* Clinically suspected UTI according to the general practitioner

Exclusion Criteria:

* Urinary catheter
* Severe urinary tract abnormality (such as cancer or strictures)
* Immunosuppression (such as chronic immunosuppressant use or AIDS)
* Dementia or any other condition (including insufficient knowledge of the German language) that could affect informed consent
* Known pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively enrolled adult non-pregnant women with a suspected uncomplicated UTI (uncomplicated is defined according to German guidelines/usual care as having no symptoms or signs of systemic illness, such as fever).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | On the 1 day of inclusion
  Sensitivity of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard) of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard)
Specificity | On the 1 day of inclusion
  Specificity of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard) of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard)
Positive predictive value | On the 1 day of inclusion
  Positive predictive value of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard) of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard)
Negative predictive value | On the 1 day of inclusion
  Negative predictive value of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard) of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard)
Positive likelihood ratio | On the 1 day of inclusion
  Positive likelihood ratio of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard) of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard)
Negative likelihood ratio | On the 1 day of inclusion
  Negative likelihood ratio of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard) of point-of-care urinalysis through Sysmex PA-100-AST vs. laboratory-based urine culture (gold standard)

OTHER OUTCOMES:
Agreement of test results for antibiotic susceptibility | On the 1 day of inclusion
  Agreement of point-of-care based with laboratory-based antibiotic susceptibility test results measured through kappa coefficients

CONTACTS AND LOCATIONS:
Overall Officials: Ildikó Gágyor, MD,Professor, Principal Investigator — University Hospital Wuerzburg
Locations (2):
- Germany (2):
  - University Hospital Wurzburg, Department of General Practice, Würzburg, Bavaria
  - University Hospital Jena, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No
Data sharing of fully anonymized individual participant data can be granted under reasonable request.

REFERENCES:
- [Background] Gagyor I, Rentzsch K, Strube-Plaschke S, Himmel W. Psychometric properties of a self-assessment questionnaire concerning symptoms and impairment in urinary tract infections: the UTI-SIQ-8. BMJ Open. 2021 Feb 15;11(2):e043328. doi: 10.1136/bmjopen-2020-043328. PMID 33589460
- [Background] Alonso-Tarres C, Benjumea Moreno C, Navarro F, Habison AC, Gonzalez-Bertran E, Blanco F, Borras J, Garrigo M, Saker J. Bacteriuria and phenotypic antimicrobial susceptibility testing in 45 min by point-of-care Sysmex PA-100 System: first clinical evaluation. Eur J Clin Microbiol Infect Dis. 2024 Aug;43(8):1533-1543. doi: 10.1007/s10096-024-04862-3. Epub 2024 Jun 3. PMID 38825624